CLINICAL TRIAL: NCT02229123
Title: Levetiracetam Efficacy and Safety as First-line Treatment of Neonatal Seizures Occuring in Hypoxic-ischemic Encephalopathy Context
Brief Title: Levetiracetam Treatment of Neonatal Seizures: Safety and Efficacy Phase II Study
Acronym: LEVNEONAT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Rennes University Hospital (Other); Amiens University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-000791-26
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Seizures
Keywords: seizures; neonates; anticonvulsant treatment; levetiracetam; hypoxic-ischemic encephalopathy; electroencephalography
MeSH Terms: conditions — Seizures; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Intervention Model Description: LEVNEONAT-1 is an open and sequential dose-finding study with 1 loading dose of 30, 40 and 50 mg/kg and 8 quarter-loading maintenance doses for a 3-day treatment. The optimal dose will be the one estimated to be associated with a toxicity not exceeding 10% and an efficacy higher than 60%. Efficacy has been defined by a seizure burden reduction of 80% after the loading dose. A 2-patient cohort will be necessary at each dose level to consider an upper dose level assignment with a dynamic consideration of each participant data. The maximal sample size expected is 30 participants patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous levetiracetam (Experimental): 1 loading dose of 30, 40 or 50 mg/kg administered intra-venously. Maintenance treatment: one intra-venous injection /8h, 8 doses in total for a 3-day treatment. Maintenance dose corresponds to the loading dose quarter i.e. 7.5, 10 or 12.5 mg/kg.
  Interventions: Drug: Intravenous Levetiracetam

INTERVENTIONS:
Drug: Intravenous Levetiracetam — Open-study. If seizure lasting more than 3 minutes on EEG recording or brief repeated seizures (more or equal to 2 seizures lasting more than 20 seconds on a 1 hour-interval), the loading-dose of LEV allocated to patient is infused followed by the 8 maintenance dose.

SUMMARY:
LEVNEONAT is a multicentre French clinical trials with the aim to develop new treatment strategies for the treatment of neonatal seizures using Levetiracetam. The purpose of this study is to determine the correct dosing, safety and efficacy for intravenous levetiracetam as first line treatment in term newborn babies with seizures in hypoxic-ischemic encephalopathy context. This new anticonvulsivant drug is a promising treatment for seizures in newborns.

DETAILED DESCRIPTION:
Article Focus

* The principal aim of LEVNEONAT-1 is to determine the levetiracetam optimal dose defined as the highest efficient dose under toxicity restrictions for treating neonatal seizures.
* LEVNEONAT-1 is an open-label, sequential dose-finding study with 3 increasing dose levels of levetiracetam.

Strenghts and limitation of study

* For the first time, levetiracetam will be used as the first-line treatment of neonatal seizures and not as an add-on therapy.
* Statistical model is designed for a rare clinical situation with a sequential adaptive method updating in real time the dose allocation for next patient by using all available data from previous participants.
* The targeted population, i.e. the newborn less than 3 days of life, is particularly sensitive and the written consent of both parents is required before the levetiracetam administration.

ELIGIBILITY:
Eligibility Criteria:

1. Male or female term baby with gestational age of 36-43 weeks and postnatal age < or= 72 hours
2. One or more of the following :

   * APGAR score < 5 at 5 mins
   * Umbilical cord or arterial blood sample (within one hour after birth): pH <7.0 or base deficit > or = 16 mmol/L or lactates > or equal to 11 mmol/L
   * Abnormal neurological examination before 6 hours of life
3. Suspected clinical or EEG seizures

Inclusion criteria:

* A seizure lasting more than 3 minutes or more than 2 seizures lasting more than 20 seconds on a 1 hour-period on standard EEG recording 4 hours before the levetiracetam loading dose
* Availability of 8 electrode EEG recording
* Written informed consent of both parents or the authorized guardians
* Subscription to social security health insurance are required

Exclusion Criteria:

* Suspected or confirmed brain malformation, inborn error of metabolism, genetic syndrome or major congenital malformation
* Congenital (in utero) infection (TORCH)
* Babies who have received phenobarbital or any other anticonvulsive medication other than a bolus of midazolam for intubation
* Anuria/renal failure defined as serum creatinine > 150 micromol/L
* Seizures secondary to treatable metabolic etiology as hypoglycemia and hypocalcemia
* Corrected QT interval (QTc) greater than 450 milliseconds on the electrocardiogram (ECG) prior to inclusion in the presence or absence of a condition that promotes QT prolongation (hypokalemia, maternal treatment during childbirth or treatment of the child with drugs known to prolong QT),
* Participation to an interventional research study

Ages: 36 Weeks to 43 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Levetiracetam Efficacy on EEG recording | the period just before the LEV loading dose (from 20 min to 3 hours) and the 3 hour time-interval from 1 hour 15 min (T11/4) to 4 hours 15 min (T41/4) after the starting of loading dose infusion (T0)
  Efficacy has been defined as an 80% reduction of seizure burden on EEG recording.
Levetiracetam Short-Term Toxicity | 6 days from the loading dose
  Short-term toxicity focuses on 4 adverse events potentially attributable to LEV occurring in the 6 days following the loading dose: i) Severe apnoea leading to mechanical ventilation during the 4-hour period following the LEV infusion; ii) Anaphylactic shock occurring during the 30 minutes following the LEV infusion; iii) Toxic epidermic necrosis; iv) Stevens-Jonhson Syndrome. Short-term toxicity has been designed to trigger quickly a decreasing dose allocation to the next potential participant through a e-CRF alert.
Levetiracetam Long-Term Toxicity | 30 days from the loading dose
  Long-term toxicity includes all the adverse events observed and declared to the pharmacovigilance unit up to the hospital discharge or the 30th day of life at the latest.

SECONDARY OUTCOMES:
Levetiracetam Elimination Clearance | at 30 min, 4 hours and 7 hours after the end of loading dose infusion, respectively and at 1 to 3 hours and 12 hours to 18 hours after the last levetiracetam maintenance dose, respectively.
  The mean values of the elimination clearance and their respective interindividual variability will be estimated.
Levetiracetam Distribution Volume | at 30 min, 4 hours and 7 hours after the end of loading dose infusion, respectively and at 1 to 3 hours and 12 hours to 18 hours after the last levetiracetam maintenance dose, respectively.
  The mean values of distribution volumes and their respective interindividual variability will be estimated.
Plasmatic Levetiracetam Maximal Concentration | 30 min, 4 hours and 7 hours after the end of Levetiracetam loading dose infusion
  Plasmatic Peak Value of Levetiracetam Loading dose will be assessed.
Levetiracetam Loading Dose Area under Curve | 30 min, 4 hours and 7 hours after the end of Levetiracetam loading dose infusion
  ndividual PK parameters will be estimated and used to calculated the AUC corresponding to the loading dose, after the first maintenance dose.
Levetiracetam Entire Treatment Area Under Curve | at 30 min, 4 hours and 7 hours after the end of loading dose infusion, respectively and at 1 to 3 hours and 12 hours to 18 hours after the last Levetiracetam maintenance dose, respectively.
  Individual PK parameters will be estimated and used to calculated the cumulative AUC of the entire treatment.
Seizure recurrence from the Efficacy criteria completion to day 6 | from 4h15 after the loading dose to 6 days
  Clinical or electric seizures recurrence after the efficacy criteria assessment and up to the complete levetiracetam elimination (estimated 5 half-life) will be reported by investigator.
Levetiracetam Efficacy according to the seizure burden intensity prior to loading dose | after the complete recruting period
  A new analysis will be performed retrospectively by adjusting the efficacy criteria to the seizure burden on the pre-treatment EEG. Two subgroups will be considered according to the seizure burden (SB) intensity on the pre-treatment EEG, i.e equal or above to 50% of the EEG recording duration (high SB group) and strictly under 50% of it (low SB group), respectively. LEV efficacy will be considered positive when a SB reduction of 50% will be observed on the post-treatment EEG recording in the high SB group whereas the reduction of 80% will be still valid for the low SB group.

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Favrais, Dr, Study Chair — University Hospital of Tours; Geraldine FAVRAIS, Dr, Principal Investigator — University hospital of Tours
Locations (8):
- France (8):
  - Service de réanimation néonatale, Angers
  - Service de réanimation néonatale, Lille
  - Service de réanimation et service néonatale, Orléans
  - Service de réanimation néonatale et pédiatrique, Paris
  - Service de réanimation néonatale, Reims
  - Néonatologie, Rennes
  - Service de Pédiatrie néonatale et réanimation, Rouen
  - Service de Néonatologie, Tours

REFERENCES:
- [Result] Favrais G, Ursino M, Mouchel C, Boivin E, Jullien V, Zohar S, Saliba E. Levetiracetam optimal dose-finding as first-line treatment for neonatal seizures occurring in the context of hypoxic-ischaemic encephalopathy (LEVNEONAT-1): study protocol of a phase II trial. BMJ Open. 2019 Jan 24;9(1):e022739. doi: 10.1136/bmjopen-2018-022739. PMID 30679288